CLINICAL TRIAL: NCT03630445
Title: Impact of Slowly Digestible Carbohydrates on Gastric Emptying Rate Suggests Activation of Ileal Brake Response
Brief Title: Slowly Digestible Carbohydrates and the Ileal Brake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: General Mills (Industry)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Distinguished Professor of Food Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1502015807
Record Dates: First submitted 2018-06-27; First posted 2018-08-14 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Appetitive Behavior
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Appetitive Behavior | interventions — Starch; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Isomaltooligosaccharides (IMOs) (Experimental): Isomaltooligosaccharides (IMOs) incorporated into a yogurt test meal.
  IMOs are a mixture of short-chain carbohydrates with a purported slow digestion property.
  Interventions: Other: Isomaltooligosaccharides (IMOs)
- Xtend® sucromalt (Experimental): Xtend® sucromalt incorporated into a yogurt test meal.
  Sucromalt is derived from a combination of sucrose (cane or beet sugar) and maltose (corn sugar), yet it has been found to be slowly digested.
  Interventions: Other: Xtend® sucromalt
- Combination of IMOs and Xtend® sucromalt (Experimental): Combination of IMOs and Xtend® sucromalt incorporated into a yogurt test meal.
  Interventions: Other: Combination of IMOs and Xtend® sucromalt
- Raw corn starch (Experimental): Raw corn starch incorporated into a yogurt test meal.
  Raw corn starch is uncooked starch from corn. Because it is not cooked, it has a slow digestion property.
  Interventions: Other: Raw corn starch
- Maltodextrin (Experimental): Maltodextrin incorporated into a yogurt test meal.
  Maltodextrin is a type of starchy carbohydrate (polysaccharide) composed of units of D-glucose (simple sugars). The maltodextrin used for this study had a fast digestion property.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: Isomaltooligosaccharides (IMOs) — Isomaltooligosaccharides (IMOs) incorporated into yogurt were tested for gastric emptying rate, glycemic response, appetitive response, and fermentability.
  Arms: Isomaltooligosaccharides (IMOs)
Other: Xtend® sucromalt — Xtend® sucromalt incorporated into yogurt was tested for gastric emptying rate, glycemic response, appetitive response, and fermentability.
  Arms: Xtend® sucromalt
Other: Combination of IMOs and Xtend® sucromalt — A combination of IMOs and Xtend® sucromalt incorporated into yogurt was tested for gastric emptying rate, glycemic response, appetitive response, and fermentability.
  Arms: Combination of IMOs and Xtend® sucromalt
Other: Raw corn starch — Raw corn starch incorporated into yogurt was tested for gastric emptying rate, glycemic response, appetitive response, and fermentability.
  Arms: Raw corn starch
Other: Maltodextrin — Maltodextrin incorporated into yogurt was tested for gastric emptying rate, glycemic response, appetitive response, and fermentability.
  Arms: Maltodextrin

SUMMARY:
The ileal brake is a feedback mechanism controlling stomach-mediated transit of a meal, for which gastric emptying can be used as an indicator. Previously, slowly digestible carbohydrates (SDCs) were shown to activate the ileal brake in a rat model; the current research aimed to determine the effect of common SDCs in humans.

DETAILED DESCRIPTION:
Diets containing slowly digestible carbohydrates (SDCs), in the form of starch-entrapped microspheres that digest into the ileum, were previously shown to reduce food intake in a diet-induced obese rat model by activating the gut-brain axis. These results suggested that SDCs trigger the ileal brake, which is a feedback mechanism controlling stomach-mediated transit of a meal. The ileal brake is characterized by delayed gastric emptying rate and increased satiety. The goal of this work was to determine if common SDCs trigger the ileal brake in humans, using gastric emptying rate as a proxy indicator. In a human study, SDCs were delivered through a semi-solid yogurt matrix, and gastric half-emptying time and postprandial glycemic response were assessed. The study was a five-arm, double-blind, crossover design with a one-week washout period between treatments (n=20, 9 females, 11 males). Four different carbohydrate ingredients (SDCs: isomalto-oligosaccharides (IMO), Xtend® sucromalt, and raw corn starch; and non-SDC: maltodextrin) were incorporated individually, or in combination, into yogurt products matched in energy density and viscosity. Participants consumed 300 g test meals of yogurt formulated with one or a combination of the carbohydrate ingredients after an overnight fast. Gastric emptying rates and glycemic response were measured using a 13C-labeled octanoic acid breath test and continuous glucose monitors, respectively. Glucose readings were continuously monitored 24 h prior to and 48 h after test meal consumption, and breath samples were collected for a 4 h period following test meal consumption.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25 kg/m2
* Stable weight for the past 3 months (i.e. +/- 2..5 kg)
* Regular eating patterns, including breakfast consumption

Exclusion Criteria:

* Gastrointestinal disease
* Smokers
* Peri- or post-menopausal women
* Celiac disease (yogurts may contain ingredients with wheat origin)
* Allergies, including dairy, lactose, and gluten
* Pregnant and lactating women
* Following a weight reduction program or having followed one during the last 3 months
* Acute or chronic disease
* Alcohol consumption > 30 units/week
* Hypertension
* Diabetes
* Previous bariatric surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rate | Acute study; 4 hours of measurement after consumption of test food
  Breath test was performed using 13C-octanoic acid mixed into test meals
Glycemic response | Acute study; 4 hours of measurement after consumption of test food
  Blood glucose was measured using a continuous glucose monitor
Appetite ratings (Visual Analog Scale, VAS) | Acute study; 4 hours of measurement after consumption of test food
  Hunger and fullness scores were measured using a 10-cm scale (0 = weakest feeling of hunger or fullness and 10 = strongest feeling of hunger or fullness) after consumption of test food. Weaker feelings of hunger and stronger feelings of fullness indicate better outcomes.

SECONDARY OUTCOMES:
Breath hydrogen (fermentability) | Acute study; 4 hours of measurement after consumption of test food
  Breath samples were collected in 15-minute intervals for 4 hours after consumption of test food and analyzed for hydrogen levels using a breath analyzer. Breath hydrogen levels are indicative of a food's fermentability.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers

REFERENCES:
- [Derived] Chegeni M, Hayes AMR, Gonzalez TD, Manderfeld MM, Lim J, Menon RS, Holschuh NM, Hedges ME, Hamaker BR. Activation of gastrointestinal ileal brake response with dietary slowly digestible carbohydrates, with no observed effect on subjective appetite, in an acute randomized, double-blind, crossover trial. Eur J Nutr. 2022 Jun;61(4):1965-1980. doi: 10.1007/s00394-021-02770-2. Epub 2022 Jan 26. PMID 35079895